CLINICAL TRIAL: NCT01870804
Title: Impact of Early High-dose Atorvastatin Versus Rosuvastatin on Contrast Induced Acute Kidney Injury in Unselected Patients With Non- ST Elevation Acute Coronary Syndromes Scheduled for Early Invasive Strategy.
Brief Title: Atorvastatin Versus Rosuvastatin on Contrast Induced Acute Kidney Injury (PRATO-ACS 2)
Acronym: PRATO-ACS-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Cardiopatici Toscani (Other)
Responsible Party: Principal Investigator, Anna Toso, MD, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 472013
Record Dates: First submitted 2013-05-30; First posted 2013-06-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Acute Coronary Syndrome
Keywords: Statins; Contrast-Induced Acute Kidney Injury; Periprocedural Myocardial Damage
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Active Comparator): Rosuvastatin (40 mg on-admission followed by 20 mg/day) until discharge; then 20 mg/day (10 mg/day if creatinine clearance < 30 ml/min)
  Interventions: Drug: Rosuvastatin
- Atorvastatin (Active Comparator): atorvastatin (80 mg on-admission followed by 40 mg/day before and after discharge)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Arms: Rosuvastatin
Drug: Atorvastatin
  Arms: Atorvastatin

SUMMARY:
The aim of the project is to compare the nephro-protective effects of high-dose atorvastatin and high-dose rosuvastatin on the incidence of Contrast Induced-Acute Kidney Injury in patients with non-ST-elevation acute coronary syndromes scheduled for early invasive strategy.

DETAILED DESCRIPTION:
This is a prospective, single-centre, randomized study, designed to compare the nephro-protective effects of high-dose atorvastatin and high-dose rosuvastatin on the incidence of Contrast Induced-Acute Kidney Injury (CI-AKI). Consecutive statin-naïve patients admitted in the investigators institution for non-ST elevation Acute Coronary Syndrome (NSTE-ACS) and scheduled for early invasive strategy will be eligible.

Patients are randomized into two groups: 1) high-dose rosuvastatin (40 mg on-admission followed by 20 mg/day); 2) high-dose atorvastatin (80 mg on-admission followed by 40 mg/day). Randomization will be performed on-admission by computerized open-label assignment in blinded envelopes used in a consecutive fashion. All patients receive the standard pre-procedural hydration. The primary end-point is the proportion of patients with an increase in serum creatinine of ≥ 0.5 mg/dl or ≥ 25% above baseline within 72 hours after contrast medium administration. The secondary end-points are persistent worsening of renal damage (eGFR reduction >= 25% at 30 days) and cumulative adverse clinical events at follow-up. Specifically: death, myocardial infarction, dialysis, stroke or persistent renal damage at 30 days; death or myocardial infarction at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive statin-naive patients with non ST-elevation acute coronary syndrome admitted to our institution and scheduled for early invasive strategy are considered for enrollment

Exclusion Criteria:

* Current statin treatment
* High-risk features warranting emergency coronary angiography (within 2 hours)
* Acute renal failure or end-stage renal failure requiring dialysis or serum creatinine ≥ 3 mg/dl
* Severe comorbidities which precluded early invasive strategy
* Contraindications to statin treatment
* Contrast media administration within the last 10 days
* Pregnancy
* Refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2013-05; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Contrast Induced-Acute Kidney Injury | 72 hours
  Increase in serum creatinine ≥ 0.5 mg/dl or ≥ 25 % within 72 hours of contrast medium exposure

SECONDARY OUTCOMES:
Renal function at 30 days | 30 days after discharge
  Estimation of the glomerular filtration rate in all patients at 30 days
Cardiovascular and renal outcome | 30 days, 6 months, 12 months
  Composite cardiovascular and renal events at follow-up including acute renal failure requiring dialysis, persistent renal damage, all-causes mortality, myocardial infarction or stroke.
Anti-inflammatory effect of rosuvastatin and atorvastatin | On admission (baseline), at discharge (after 5 days) & at 30 days
  High-sensitivity C-reactive protein (hs-CRP)will be measured on admission, at discharge and at 30 days.
Lipid-modulatory effects of atorvastatin and rosuvastatin | On admission (baseline), at discharge (after 5 days) & at 30 days
  Low density lipoprotein (LDL) levels will be determined on admission, at discharge and at 30 days.
Myocardial Damage | During hospitalization (average 5 days)
  Total cardiac biomarkers release during the index event

CONTACTS AND LOCATIONS:
Overall Officials: Anna Toso, MD, Principal Investigator — Prato Hospital, Italy
Locations (1):
- Cardiology Division, Prato Hospital, Prato, Prato, Italy

REFERENCES:
- [Derived] Toso A, Leoncini M, Maioli M, Tropeano F, Villani S, Bellandi F. A Prospective, Randomized, Open-Label Trial of Atorvastatin versus Rosuvastatin in the Prevention of Contrast-Induced Acute Kidney Injury, Worsened Renal Function at 30 Days, and Clinical Events After Acute Coronary Angiography: the PRATO-ACS-2 Study. Cardiorenal Med. 2020;10(5):288-301. doi: 10.1159/000506857. Epub 2020 May 20. PMID 32434204